CLINICAL TRIAL: NCT06404710
Title: Effects of Progressive Muscle Relaxation Exercises Applied After Heart Surgery on Anxiety, Pain, Sleep and Effect on Healing Quality
Brief Title: Progressive Muscle Relaxation Exercise Applied After Heart Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Çığla Arslankılıç, Registered nurse, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/26
Record Dates: First submitted 2024-04-30; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: the Participant Wishes to Leave the Study
Keywords: progressive muscle relaxation; anxiety; quality of recovery; heart surgery; sleep; pain
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled (experimental and control group)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Scales will be filled in for the control group without any progressive relaxation exercise.
- Exercise (Experimental): Scales will be filled in by the intervention group by performing a progressive relaxation exercise.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Participants in this group will be given a gradual muscle relaxation exercise.
  Arms: Exercise

SUMMARY:
Various methods are used to prolong life and improve quality of life in heart diseases.

There are surgical treatment options. Heart surgery is a major surgery and surgery Due to common postoperative symptoms, follow-up and follow-up in the early postoperative period maintenance is important.Progressive relaxation exercise; optimization of analgesia, pain management, reduction of side effects, regulation of vital signs, increase in sleep qualityIt has been reported that it provides positive effects on many systems and increases the success of the surgical process. It has been stated in research that it can increase.In this study, patients who had undergone cardiac surgery and were treated as inpatients progressive muscle relaxation in reducing pain, reducing anxiety, and improving the quality of sleep and recovery It was aimed to determine the effect of the exercises.

DETAILED DESCRIPTION:
In the literature reviews, it has been determined that the treatment applied to patients after cardiac surgery. A study examining the effects of progressive muscle relaxation exercise on pain, sleep and recovery quality. No study was found. This study shows that progressive muscle relaxation exercise affects pain, sleep and Its effect on the quality of recovery will be evaluated. Progressive muscle relaxation after heart surgery. If the exercises are found to be effective, they should be implemented routinely in the surgical ward. will be recommended. With this study, cardiac surgery is included in the literature in the field of surgical nursing.

The application of progressive muscle relaxation exercises after surgery has a significant effect on pain, recovery quality andIt is aimed to contribute with findings regarding its effect on sleep quality. of nurses using nonpharmacological methods in clinics; professional of the nursing profession It will increase their practice, independent role and quality of care. After heart surgery. Reducing postoperative pain and anxiety with progressive muscle relaxation exercises, It is thought that it may be useful in improving sleep quality and recovery quality.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study,
* Those who are 18 years of age and over,
* Those who underwent coronary bypass graft surgery
* Communication difficulties and mental disability regarding vision, hearing and speech non,
* Blood pressure measurement does not need to be done on an outpatient basis,
* Any postoperative complications (bleeding, nausea, vomiting, etc.) not occurring,
* Analgesic medication should be administered before the first intervention planned to be performed after the surgery.

not implemented,

* Any medication etc. without substance addiction,
* Does not have chronic pain in any part of the body,
* Those who were extubated after cardiac surgery and were not given sedating medication
* All non-pregnant patients will be included in the sample.

Exclusion Criteria:

• Any symptoms such as severe bleeding, nausea or vomiting after the surgical procedure.

developing complications,

* Patient-controlled analgesia (PCA) for pain control after surgery applied
* Those with deformity in the chest area,
* Preoperative respiratory function test is not within normal limits,
* Patients with Chronic Obstructive Pulmonary Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
NUMERICAL RATING SCALE | First day before surgery, first 4 days after surgery and 20 days after discharge
  This scale contains numbers from 1 to 10. 1: not at all, 10: very much. Patients' pain will be measured.
VISUAL COMPARISON SLEEP SCALE | 3rd day after surgery and 20 days after discharge
  Each item in the scale is evaluated using a visual comparison technique on a graph between 0 (left end) and 100 (right end), the minimum score that can be obtained from the scale is 0 and the maximum score is 1000. An increase in the score obtained from the scale indicates that sleep quality decreases. It consists of 15 items in total.
State Anxiety Scale | 3rd day after surgery and 20 days after discharge
  Anxiety level is scored as "(1) not at all, (2) a little, (3) a lot and (4) completely". The scores obtained from the scale theoretically range between 20 and 80. A high score indicates a high level of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Özel Bilgi Hastanesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided